CLINICAL TRIAL: NCT04037657
Title: A Phase 1b, Positive-controlled, Dose-escalation Study to Determine the Safety, Pharmacodynamics and Pharmacokinetics of a Single Intravenous Dose of HSK3486 in Healthy Female Subjects.
Brief Title: Evaluating the Safety, Pharmacodynamics and Pharmacokinetics of HSK3486 in Healthy Female Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK3486-Australian-02
Record Dates: First submitted 2019-07-20; First posted 2019-07-30 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2015-12

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): 0.288 mg/kg ，0.432 mg/kg ，0.540 mg/kg ，0.648 mg/kg，0.810 mg/kg There were five cohorts of six subjects per cohort (5 HSK3486:1 propofol).
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): 2.5 mg propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — HSK3486 was administered as a single dose over a 1 minute infusion period. There were five cohorts of six subjects per cohort (5 HSK3486:1 propofol).
  Arms: HSK3486
Drug: Propofol — Propofol, at a dose of 2.5 mg/kg, was administered as a 1 minute infusion at a constant rate via infusion pump.
  Arms: Propofol

SUMMARY:
This study was a single-center positive-controlled, randomized, dose-escalation study of HSK3486 in healthy female subjects administered as a single IV bolus dose.Subjects were confined to the study unit from the evening of Day -1 until the morning of Day 2, then were required to return for a follow up visit on Day 5. Intensive safety, PD and PK assessments were performed prior to dosing on Day 1 until 24 hours post-dose (Day 2).

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 - 49 years (inclusive)
* Women of child-bearing potential agreed to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy
* Negative serum pregnancy test
* In general good health without CS medical history
* American Society of Anesthesiologists (ASA) Physical Status Classification of I or II
* Body Mass Index (BMI) between 18 and 30 kg/m2 (inclusive)
* Negative screen for drugs of abuse, alcohol, hepatitis B surface antigen (HBs-Ag), hepatitis C virus antibody (HCV-Ab) and Human Immunodeficiency Virus (HIV) at screening; and drugs of abuse, alcohol pre dose on Day -1
* Normal or non-CS findings on a physical examination, 12-lead Electrocardiogram (ECG) and vital signs (respiratory rate between 12 and 20 breaths per minute, blood pressure (BP) between 100-140/60-90 mmHg, heart rate between 50-99 beats per minute, temperature between 35.8°C and 37.5°C and pulse oximetry values > 95% on room air)
* Clinical laboratory values within the normal limits as defined by the clinical laboratory, unless the PI decided that out-of-range values were not CS
* Able to provide written informed consent
* Willing and able to follow study instructions and likely to complete all study requirements
* Suitable venous and arterial access

Exclusion Criteria:

* History of allergy or sensitivity to: propofol, components of Fresofol 1% MCT/LCT propofol, or HSK3486 (excipients soy bean oil, glycerine, triglycerides, purified egg phospholipids, sodium oleate and sodium hydroxide), or plain lignocaine
* History of CS problems with general anesthesia
* Current smoker, or a history of regular (more than weekly) use of tobacco- or nicotine-containing products within 2 months prior to screening
* History of excessive alcohol intake (more than four standard drinks daily, on average) or use of recreational drugs within the last 3 months CONFIDENTIAL HSK3486 SAD_02 Sichuan Haisco Pharmaceutical Co., Ltd Version: 13 Nov 2015 Page 19 of 513
* Use of prescription or over the counter medications within 7 days of Investigational Product administration, with the exception of contraceptive medications, paracetamol, oral non-steroidal anti-inflammatory agents, topical over the counter preparations and routine vitamins (if they do not exceed an intake of 20 to 600 times the recommended daily dose), unless agreed as non-clinically relevant by the PI and Sponsor.
* Standard donation of blood within 30 days of the study
* Donation of plasma or participation in a plasmapheresis program within 7 days preceding this study
* Receipt of any investigational study drug within 30 days prior to screening
* Unable to fast for the 6 hours prior to Investigational Product administration
* CS (as judged by the Investigator) presence of acute illness (e.g. gastrointestinal illness, infection such as influenza, upper respiratory tract infection) at admission to the clinical study unit
* Anticipated need for surgery or hospitalization during the study
* Anatomical abnormality that would potentially interfere with airway management under unconscious sedation or anesthesia
* History of posture-related gastric reflux more than twice weekly
* History of seizures or epilepsy
* History of ischaemic heart disease
* History of brady- or tachy-dysrhythmias requiring medical care
* History of asthma, with bronchospasm requiring treatment in the last 3 months
* Any condition, which in the Investigator's opinion, puts the subject at significant risk, could confound the study results or may interfere significantly with the subject's participation in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2015-11-13 (Actual)

PRIMARY OUTCOMES:
Safety by measurement of Adverse Events | First dose of study drug on day 1
Bispectral index （BIS） | From first dose of study drug until fully alert on day 1
Modified observer's assessment of alertness/sedation（MOAA/S） | Time Frame: From first dose of study drug until fully alert on day 1
  Observe the change of modified observer's assessment of alert /sedation during the whole trial

SECONDARY OUTCOMES:
Median effective dose (ED50) | From first dose of study drug until fully alert on day 1
Peak concentration (Cmax) | From the start of administration to 48 hours after administration
Time to plasma peak concentration(Tmax) | From the start of administration to 48 hours after administration
Area Under the Curve (AUC0-30min, AUC0-1h, AUC0-last, and AUC0-inf) | From the start of administration to 48 hours after administration
Total clearance (CL) | From the start of administration to 48 hours after administration

IPD SHARING:
Plan to Share IPD: Undecided